CLINICAL TRIAL: NCT04674891
Title: Effects of Cervical Stabilization Exercises on Respiratory Strength in Chronic Neck Pain Patients With Forward Head Posture
Brief Title: Cervical Stabilization Exercises on Respiratory Strength in Chronic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/LHR/20/1048 Tooba Arif
Record Dates: First submitted 2020-12-16; First posted 2020-12-19 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2021-03

CONDITIONS: Neck Pain
Keywords: NDI, NPRS, CVA, SBC
MeSH Terms: conditions — Neck Pain; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- baseline physical therapy treatment (Active Comparator): baseline physical therapy treatment ,Control group- Group A
  Interventions: Other: baseline physical therapy treatment
- Cervical Stabilization exercises (Experimental): baseline physical therapy treatment along with Cervical Stabilization exercises- Experimental Group- Group B
  Interventions: Other: Cervical Stabilization exercises

INTERVENTIONS:
Other: baseline physical therapy treatment — Group A was control group and the patients received Conventional treatment protocol for 4 weeks which included 3 sessions per week. Patients received hot pack for 15 min and TENS (Transcutaneous Electric Nerve Stimulation) for 10 min. After that Cervical isometric exercises will be performed in sitting (10sec hold,10 to 15 reps)
  Arms: baseline physical therapy treatment
Other: Cervical Stabilization exercises — Group B was experimental group and received baseline physiotherapy treatment in addition to Cervical Stabilization exercises. Pillow was placed beneath cervical spine in supine position and guided patients to nod head as though they said 'yes' and asked them to hold for 10 seconds. 10 repetitions were done before progressing to the next target level.
  4 weeks (3 sessions per week)
  * Hot pack: 10 min
  * TENS: 10 min
  * Cervical isometric exercises in sitting (10sec hold,10 to 15 reps)
  * Cervical Stabilization exercises (10 sec hold, 10 reps)
  On eligible participants baseline assessment was taken on day 1, post intervention assessment was taken at the end of 4th week.
  Arms: Cervical Stabilization exercises

SUMMARY:
This project was a Randomized control trial conducted to check the effects of Cervical Stabilization Exercises on Respiratory Strength in Chronic Neck Pain Patients with Forward Head Posture, duration of study was of 6 months, convenient sampling was done, subject following eligibility criteria from Jinnah Hospital Lahore, were randomly allocated in two groups via lottery method, baseline assessment was done, Group A participants were given baseline treatment protocol for 4 weeks which included 3 sessions per week. Heating Pad applied for 15 min and TENS (Transcutaneous Electric Nerve Stimulation) for 10 min. After that Cervical isometric exercises performed in sitting (10sec hold, 10 to 15 reps). Group B was experimental group and participants were given baseline treatment in addition to Cervical Stabilization exercises for 4 weeks which included 3 sessions per week. The baseline measurement was taken on day one for Numeric Pain Rating Scale (NRPS) and Neck Disability Index (NDI). Forward head posture assessed by measuring Cranio Vertebral Angle (CVA). Respiratory muscle strengths measured by Spirometer and SBC (single breath count). All the measurements repeated at the end of fourth week. Data was analyzed by using SPSS version 20.

DETAILED DESCRIPTION:
Extensive usage of electronic gadgets in today's life leads to the musculoskeletal problems among which neck pain is the most common problem reported to physicians, orthopedics and physical therapists. Even before reporting to clinics there is long history of using over the counter pain killers. Pain avoidance behaviors let the cervical spine stiff so much that a clinician help is sought. There is huge literature regarding the management of chronic neck pain and yet after the decades of research there are gaps in treatment options. In modern age of health care, it is common goal of every healthcare to make patient self-sufficient as early as possible. The self-care models have tremendous advantages. The current study has compared the effects of cervical stabilization exercises and isometric exercises. The current study was novel in a way that there is limited literature about treating Chronic Neck Pain Patients with effects of physiotherapy on respiratory strength in improving forward head posture. All the methods were employed to see if they improve ranges along with accompanying pain and disability.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic neck pain for more than 3 months.
* Mild neck disability (NDI score 5-15)

Exclusion Criteria:

* Neck pain secondary to trauma
* Deformities of thoracic region or vertebral column
* History of any thoracic or vertebral column surgery.
* History of smoking
* Patients with any other serious pathology/red flags

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2020-03-30 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2021-01-30 (Actual)

PRIMARY OUTCOMES:
Numeric Pain rating scale | 4th week
  The NPRS is the segmented numeric version of visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of pain. The common format is a horizontal bar or line. Similar to VAS, the NPRS is anchored by terms describing pain severity extremes.

SECONDARY OUTCOMES:
Neck disability Index | 4th Week
  Methods of assessment for such disability, especially those targeted at activities of daily living which are most affected by neck pain, questionnaire 10-item scaled entitled the Neck Disability Index (NDI)

OTHER OUTCOMES:
Spirometer | 4th Week
  A spirometer is an apparatus for measuring the volume of air inspired and expired by the lungs. A spirometer measures ventilation, the movement of air into and out of the lungs. The spirogram will identify two different types of abnormal ventilation patterns, obstructive and restrictive
Single Breath Count( SBC) | 4th Week
  To perform, ask patient to count out loud after maximal inspiration. Ability to reach 50 indicates normal respiratory function. Single breath count of less than 15 typically correlates with low forced vital capacity (FVC) and respiratory muscle weakness

CONTACTS AND LOCATIONS:
Overall Officials: Syed Shakil Ur Rehman, Principal Investigator — Riphah International University
Locations (1):
- Jinnah Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Miranda IF, Wagner Neto ES, Dhein W, Brodt GA, Loss JF. Individuals With Chronic Neck Pain Have Lower Neck Strength Than Healthy Controls: A Systematic Review With Meta-Analysis. J Manipulative Physiol Ther. 2019 Oct;42(8):608-622. doi: 10.1016/j.jmpt.2018.12.008. Epub 2019 Nov 23. PMID 31771837
- [Background] Migliarese S, White E. Review of Forward-Head Posture and Vestibular Deficits in Older Adults. Current Geriatrics Reports. 2019;8(3):194-201.
- [Background] Gurudut P, Welling A, Chodankar A. Effect of self-care exercises in forward head posture on craniovertebral angle and craniocervical flexion endurance: A pilot study. Indian Journal of Physical Therapy and Research. 2020;2(1):25.
- [Background] Son K-k, Cynn H-S, Lee J-H, Park D-H, Kim B-B. Effects of Deep Cervical Flexor Exercise with Visual Guide on Muscle Activity and Craniovertebral Angle in Subjects with Forward Head Posture. Korean Society of Physical Medicine. 2019;14(2):53-61.
- [Background] Koseki T, Kakizaki F, Hayashi S, Nishida N, Itoh M. Effect of forward head posture on thoracic shape and respiratory function. J Phys Ther Sci. 2019 Jan;31(1):63-68. doi: 10.1589/jpts.31.63. Epub 2019 Jan 10. PMID 30774207
- [Background] Mathur H, Khan SA, Siddiqui ZA. Effect of forward head posture on swallowing: Review of Literature. 2019
- [Background] Herman PM, Vernon H, Hurwitz EL, Shekelle PG, Whitley MD, Coulter ID. Clinical Scenarios for Which Cervical Mobilization and Manipulation Are Considered by an Expert Panel to Be Appropriate (and Inappropriate) for Patients With Chronic Neck Pain. Clin J Pain. 2020 Apr;36(4):273-280. doi: 10.1097/AJP.0000000000000800. PMID 31985500
- [Background] Alsultan F, De Nunzio AM, Rushton A, Heneghan NR, Falla D. Variability of neck and trunk movement during single- and dual-task gait in people with chronic neck pain. Clin Biomech (Bristol). 2020 Feb;72:31-36. doi: 10.1016/j.clinbiomech.2019.11.019. Epub 2019 Nov 28. PMID 31809920
- [Background] Storto CJ, Garcez AS, Suzuki H, Cusmanich KG, Elkenawy I, Moon W, Suzuki SS. Assessment of respiratory muscle strength and airflow before and after microimplant-assisted rapid palatal expansion. Angle Orthod. 2019 Sep;89(5):713-720. doi: 10.2319/070518-504.1. Epub 2019 Mar 21. PMID 30896250
- [Background] Kalita J, Kumar M, Misra UK. Serial single breath count is a reliable tool for monitoring respiratory functions in Guillain-Barre Syndrome. J Clin Neurosci. 2020 Feb;72:50-56. doi: 10.1016/j.jocn.2020.01.032. Epub 2020 Jan 22. PMID 31982274
- [Background] Uysal SC, Tuzun EH, Eker L, Angin E. Effectiveness of the muscle energy technique on respiratory muscle strength and endurance in patients with fibromyalgia. J Back Musculoskelet Rehabil. 2019;32(3):411-419. doi: 10.3233/BMR-181287. PMID 30475751
- [Background] Pawaria S, SuDhan DS, Kalra S. Effectiveness of Cervical Stabilisation Exercises on Respiratory Strength in Chronic Neck Pain Patients with Forward Head Posture-A Pilot Study. Journal of Clinical and Diagnostic Research. 2019;13(4).
- [Background] Lee H-j, Park H-s, Park J-m. The Effects of Cervical Stabilization Exercise on Neck Pain, Range of Motion, and Deep Cervical Muscle Strength in Patients With Chronic Neck Pain. The Journal of Korean Academy of Orthopedic Manual Physical Therapy. 2019;25(1):9-19
- [Background] Lee MH, Jang SH. The effects of the neck stabilization exercise on the muscle activity of trunk respiratory muscles and maximum voluntary ventilation of chronic stroke patients. J Back Musculoskelet Rehabil. 2019;32(6):863-868. doi: 10.3233/BMR-170839. PMID 30958329
- [Background] Kim G-C, HwangBo P-N. Effects of cervical stabilization exercise using pressure biofeedback on neck pain, forward head posture and acoustic characteristics of chronic neck pain patients with forward head posture. Korean Society of Physical Medicine. 2019;14(1):121-9.
- [Background] Young IA PT, DSc, Dunning J PT, DPT, Butts R PT, PhD, Mourad F PT, DPT, Cleland JA PT, PhD. Reliability, construct validity, and responsiveness of the neck disability index and numeric pain rating scale in patients with mechanical neck pain without upper extremity symptoms. Physiother Theory Pract. 2019 Dec;35(12):1328-1335. doi: 10.1080/09593985.2018.1471763. Epub 2018 Jun 1. PMID 29856244